CLINICAL TRIAL: NCT03303677
Title: Comparison of Post op Outcomes in Endoscopic Sinus Surgery Using Varying Nasal Sinus Irrigations. Saline vs. Saline and Budesonide vs Saline, Budesonide, and Culture Directed Topical Antibiotics
Brief Title: Comparison of Topical Therapies in Post op Endoscopic Sinus Surgery Patients
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Withdrawn by sponsor
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201701952
Record Dates: First submitted 2017-09-26; First posted 2017-10-06 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Chronic Rhinosinusitis (Diagnosis)
Keywords: endoscopic sinus surgery; topical nasal therapy
MeSH Terms: conditions — Disease | interventions — Sodium Chloride; Anti-Infective Agents; Pharmaceutical Preparations; Levofloxacin; Vancomycin; Gentamicins; Ciprofloxacin; Mupirocin; Trimethoprim; Sulfamethoxazole

STUDY DESIGN:
Intervention Model Description: Randomization into one of three treatment arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Saline (Active Comparator): Post operative endoscopic sinus surgery patients using Saline nasal sinus irrigations to be performed twice daily. All patients will begin with normal saline irrigations immediately following surgery as per our department's standard of care. At their first one week post op appointment they will then begin treatment per the treatment arm.
  Interventions: Drug: Saline Nasal
- Saline and budesonide (Experimental): Post operative endoscopic sinus surgery patients using saline + budesonide nasal sinus irrigations to be performed twice daily. All patients will begin with normal saline irrigations immediately following surgery as per our department's standard of care. At their first one week post op appointment they will then begin treatment per the treatment arm.
  Interventions: Drug: Saline Nasal; Drug: Budesonide Nasal
- saline, budesonide, and topical antibiotic (Experimental): Post operative endoscopic sinus surgery patients using saline + budesonide + topical antibiotic nasal sinus irrigations. The antibiotic would be chosen based on intra operative culture sensitives as is our standard practice. The antibiotic would be selected from Levaquin, Vancomycin, Gentamicin, Ciprofloxacin, Mupirocin, and Trimethoprim/Sulfamethoxazole. All patients will begin with normal saline irrigations immediately following surgery as per our department's standard of care. At their first one week post op appointment they will then begin treatment per the treatment arm.
  Interventions: Drug: Saline Nasal; Drug: Budesonide Nasal; Drug: Topical Antibacterial (Product)

INTERVENTIONS:
Drug: Saline Nasal — topical nasal saline rinses
Drug: Budesonide Nasal — saline + budesonide nasal saline irrigation
  Arms: Saline and budesonide; saline, budesonide, and topical antibiotic
Drug: Topical Antibacterial (Product) — The antibiotic would be chosen based on intra operative culture sensitives as is our standard practice. The antibiotic would be selected from Levaquin, Vancomycin, Gentamicin, Ciprofloxacin, Mupirocin, and Trimethoprim/Sulfamethoxazole
  Other Names: Levaquin, Vancomycin, Gentamicin, Ciprofloxacin, Mupirocin, and Trimethoprim/Sulfamethoxazole
  Arms: saline, budesonide, and topical antibiotic

SUMMARY:
The goal of the study is to compare postoperative symptom scores and endoscopy findings between in patients who receive either nasal saline rinses, saline + budesonide, and saline + topical antibiotics and budesonide following endoscopic sinus surgery.

DETAILED DESCRIPTION:
The group of patients from which the study tem will recruit consists of patients referred to the University of Florida tertiary referral rhinology practice of Dr. Jeb Justice and Dr. William Collins. Patients with CRS defined by symptom, endoscopic, and radiographic criteria who are candidates for surgical intervention will be identified by the above-mentioned investigators. As part of their initial pre operative work up they will be asked to fill out SNOT-22 and RSDI surveys. As part of their surgery intraoperative cultures will be obtained from the surgically opened sinus cavities. The above radiologic, endoscopic procedures, cultures and QOL/symptoms surveys are typical in the workup of patients who present with rhinologic related problems. None of the above tests will be undertaken for the sole purpose of this study.

If the patient meets criteria, he/she will be approached by one of the investigators about participating in the research study. Information regarding the study, including the informed consent form, will be extensively discussed. If the patient agrees to take part in this study, the consent form will be provided for review and will then be signed. This consent form will be kept in a secure locked location with access given only to study staff identified in the Institutional Review Board (IRB) protocol. It will be explained to the patients that there is no obligation for them to participate in the study and that they can drop out of the study at any time without repercussions regarding their care.

If a patient elects to be a part of the study they will be randomized into one of three treatment arms. This process will be done by placing an equal number of note cards in envelopes. The note cards will contain either a "1", "2", or "3" to represent the different treatment arms. These will be placed in the envelopes, shuffled, and kept in a box in the otolaryngology clinic. At the patient's first postoperative appointment an envelope is drawn and it is documented which treatment arm the patient will be treated under.

All patients will begin with normal saline irrigations immediately following surgery as per our department's standard of care. At their first one week post op appointment they will then begin treatment per the treatment arm. The first treatment arm will consist of patients that are given only saline nasal irrigations to be performed twice daily. The second arm will be given a prescription for nasal saline + budesonide to be performed twice daily. The final arm will be given a prescription for nasal saline + budesonide + a culture directed topical antibiotic. These treatments are commonly used in our practice and will be obtained through the compounding pharmacies that are already in use by our practice.

Patients will be seen in follow up at 1-2 week, 3-4 week, 6-8 week, and 10-12 week follow up appointments. At each of these appointments they will undergo nasal endoscopy and debridement as is standard following endoscopic sinus surgery. They will also be asked to fill out SNOT-22 and RSDI surveys to monitor their progression.

The RSDI contains 30 questions designed to measure the patient's disease-specific status in the physical, emotional, and functional domains. The questions present the patient with symptoms and ask if there experience the symptoms never, almost never, sometimes, almost always, and always. These are scored as 0-4, with never getting a score of 0 and always getting a score of 4 for a total score range of 0-120.

The Snot-22 contains 22 questions with a each question scored on a visual analog scale of 1-5 where 1 represents no problems with the symptom and 5 represents the symptom is as bad as it possibly can be. The Snot-22 has a cumulative score of 0-110.

Endoscopy findings will be scored using the Lund-Kennedy endoscopy scoring system. This system grades the endoscopic findings within the paranasal sinuses for the presence of: polyps, discharge, edema, scarring and crusting . Each side of the nasal cavity is scored separately and then combined for the total score. Polyps are scored as absent (0), present in middle meatus (1), or extending beyond middle meatus (2). Discharge is scored as absent (0), thin (1), and thick or purulent (2). Scarring, crusting, and edema are each scored separately as absent (0), mild (1), or severe (2). Combing the scores from both sides of the nasal cavity a total score from 0-20 is found.

Final data will compare the pre and postoperative SNOT-22 and RSDI surveys, endoscopy findings, need for oral antibiotics, and need for oral steroids for the three treatment arms.

Cultures will be obtained for all patients during endoscopic sinus surgery as is our standard practice. During treatment patients will be treated as per standard which could include the use of oral antibiotics, oral steroids, or nasal steroid sprays as their medical condition warrants.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Chronic rhinosinusitis (CRS) defined by symptom, endoscopic, and radiographic criteria who are undergoing endoscopic sinus surgery

Exclusion Criteria:

* Age <18
* endoscopic sinus surgery for reason other than CRS

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2018-11-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in symptom scores on Sino-nasal Outcome Test (SNOT)-22 surveys | Up to 12 weeks post op
  The Snot-22 contains 22 questions with a each question scored on a visual analog scale of 1-5 where 1 represents no problems with the symptom and 5 represents the symptom is as bad as it possibly can be. The Snot-22 has a cumulative score of 0-110.
Change in symptom scores on Rhinosinusitis Disability Index (RSDI) | Up to 12 weeks post op
  The RSDI contains 30 questions designed to measure the patient's disease-specific status in the physical, emotional, and functional domains. The questions present the patient with symptoms and ask if there experience the symptoms never, almost never, sometimes, almost always, and always. These are scored as 0-4, with never getting a score of 0 and always getting a score of 4 for a total score range of 0-120.
Nasal endoscopy findings | Up to 12 weeks post op
  Lund-Kennedy endoscopy scoring system. This system grades the endoscopic findings within the paranasal sinuses for the presence of: polyps, discharge, edema, scarring and crusting. Each side of the nasal cavity is scored separately and then combined for the total score. Polyps are scored as absent (0), present in middle meatus (1), or extending beyond middle meatus (2). Discharge is scored as absent (0), thin (1), and thick or purulent (2). Scarring, crusting, and edema are each scored separately as absent (0), mild (1), or severe (2). Combing the scores from both sides of the nasal cavity a total score from 0-20 is found

CONTACTS AND LOCATIONS:
Overall Officials: Jeb Justice, MD, Principal Investigator — University of Florida
Locations (1):
- Univeristy of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rosenfeld RM, Piccirillo JF, Chandrasekhar SS, Brook I, Ashok Kumar K, Kramper M, Orlandi RR, Palmer JN, Patel ZM, Peters A, Walsh SA, Corrigan MD. Clinical practice guideline (update): adult sinusitis. Otolaryngol Head Neck Surg. 2015 Apr;152(2 Suppl):S1-S39. doi: 10.1177/0194599815572097. PMID 25832968
- [Result] Rawal RB, Deal AM, Ebert CS Jr, Dhandha VH, Mitchell CA, Hang AX, Gore MR, Senior BA, Zanation AM. Post-operative budesonide irrigations for patients with polyposis: a blinded, randomized controlled trial. Rhinology. 2015 Sep;53(3):227-34. doi: 10.4193/Rhino14.196. PMID 26363164
- [Result] Lee VS, Davis GE. Culture-directed topical antibiotic treatment for chronic rhinosinusitis. Am J Rhinol Allergy. 2016 Nov 1;30(6):414-417. doi: 10.2500/ajra.2016.30.4380. PMID 28124652
- [Result] Lim M, Citardi MJ, Leong JL. Topical antimicrobials in the management of chronic rhinosinusitis: a systematic review. Am J Rhinol. 2008 Jul-Aug;22(4):381-9. doi: 10.2500/ajr.2008.22.3189. PMID 18702902
- [Result] Rudmik L, Smith TL. Evidence-based practice: postoperative care in endoscopic sinus surgery. Otolaryngol Clin North Am. 2012 Oct;45(5):1019-32. doi: 10.1016/j.otc.2012.06.006. PMID 22980682
- [Result] Portela RA, Hootnick J, McGinn J. Perioperative care in functional endoscopic sinus surgery: a survey study. Int Forum Allergy Rhinol. 2012 Jan-Feb;2(1):27-33. doi: 10.1002/alr.20098. Epub 2011 Oct 24. PMID 22311838
- [Result] Kim ST, Sung UH, Jung JH, Paik JY, Woo JH, Cha HE, Kang IG. The effect of maxillary sinus irrigation on early prognostic factors after endoscopic sinus surgery: a preliminary study. Am J Rhinol Allergy. 2013 Sep-Oct;27(5):e158-61. doi: 10.2500/ajra.2013.27.3967. PMID 24119597
- [Result] Giotakis AI, Karow EM, Scheithauer MO, Weber R, Riechelmann H. Saline irrigations following sinus surgery - a controlled, single blinded, randomized trial. Rhinology. 2016 Dec 1;54(4):302-310. doi: 10.4193/Rhino16.026. PMID 27556896
- [Result] Kang TW, Chung JH, Cho SH, Lee SH, Kim KR, Jeong JH. The Effectiveness of Budesonide Nasal Irrigation After Endoscopic Sinus Surgery in Chronic Rhinosinusitis With Asthma. Clin Exp Otorhinolaryngol. 2017 Mar;10(1):91-96. doi: 10.21053/ceo.2016.00220. Epub 2016 Jul 21. PMID 27440128
- [Result] Jang DW, Lachanas VA, Segel J, Kountakis SE. Budesonide nasal irrigations in the postoperative management of chronic rhinosinusitis. Int Forum Allergy Rhinol. 2013 Sep;3(9):708-11. doi: 10.1002/alr.21189. Epub 2013 Jun 17. PMID 23776108
- [Result] Oakley GM, Harvey RJ. Topical Steroids. Adv Otorhinolaryngol. 2016;79:121-30. doi: 10.1159/000445148. Epub 2016 Jul 28. PMID 27466854
- [Result] Wong KK, Marglani O, Westerberg BD, Javer AR. Systemic absorption of topical gentamicin sinus irrigation. J Otolaryngol Head Neck Surg. 2008 Jun;37(3):395-8. PMID 19128645